CLINICAL TRIAL: NCT04123600
Title: Origin Stem and Logical Cup Post Market Clinical Follow-up
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Signature Orthopaedics (Industry)
Collaborators: The Cleveland Clinic (Other)
Responsible Party: Sponsor
Other Study IDs: 111-201-352
Record Dates: First submitted 2019-10-08; First posted 2019-10-11 (Actual); Last update posted 2021-09-22 (Actual); Status verified 2021-09

CONDITIONS: Hip Disease
Keywords: Hip Replacement

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Device: Origin Stem and Logical Cup — The Origin Stem is a straight, tapered, HA coated cementless femoral stem, and the Logical Cup is a porous coated acetabular cup mated with a cross-linked polyethylene liner. The components are used as part of a total joint replacement prosthesis.

SUMMARY:
The aim of the study is to monitor the performance of the Signature Orthopaedics Origin Stem and Logical Acetabular Cup as part of post-market vigilance and continuous improvement efforts.

DETAILED DESCRIPTION:
The objective of this PMCF study is to collect data confirming safety, performance and clinical benefits of the Origin Stem and Logical Cup when used for primary total hip arthroplasty at 2 years follow-up. This prospective follow-up series is necessary to obtain data specific to the Origin Stem and Logical Cup considering their relatively recent launch to the market.

The study includes pre-operative, operative, discharge, 1 year post-operative and 2 year post-operative evaluations, where data concerning the performance and safety of the device are gathered. In particular, the revision rate of the components will be monitored as the primary objective, along with pre- and post-operative measurement of the Oxford Hip Score (OHS) patient-reported outcome measure (PROM) to quantify patient satisfaction, and radiographic analysis to monitor bony response to the implant and qualify the effectiveness of the cementless fixation.

ELIGIBILITY:
Inclusion Criteria:

* patient requires unilateral primary total hip arthroplasty due to non-inflammatory degenerative joint disease (e.g. osteoarthritis, traumatic arthritis, avascular necrosis, dysplasia/DDH)
* patient must be a candidate for use of the products studied, as determined jointly by the surgeon and patient
* male and non-pregnant female patients aged 18-75
* patients who understand the conditions of the clinical evaluation and are willing to participate for the length of the prescribed follow-up

Exclusion Criteria:

* patient has active infection or sepsis (treated or untreated)
* patient has any vascular insufficiency, muscular atrophy, or neuromuscular disease severe enough to compromise implant stability or postoperative recovery.
* patient is female of child-bearing age and not taking contraceptive precautions
* patient has inadequate bone stock to support the device (e.g. severe osteopenia, family history of severe osteoporosis or osteopenia)
* patient has inflammatory joint disease (e.g. rheumatoid arthritis)
* patient has known moderate to severe renal deficiency
* patient has a known or suspected metal sensitivity
* patient is immuno-suppressed with diseases such as AIDS or is receiving high dose of corticosteroids
* patient has an emotional or neurological condition that would pre-empt their ability or unwillingness to participate in the clinical evaluation including mental illness, mental retardation or drug abuse
* patient is severely overweight with a BMI>40.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients of the Cleveland Clinic
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2019-11-19 (Actual); Primary Completion 2023-11-19 (Estimated); Study Completion 2023-11-19 (Estimated)

PRIMARY OUTCOMES:
Stem and Cup Survival Rate | up to 2 years
  The implant survival rate based on removal of the device for any reason as determined following the Kaplan-Meier method.

SECONDARY OUTCOMES:
Oxford Hip Score (OHS) | up to 2 years
  The OHS is a patient reported outcome measure (PROM) used to quantify patient satisfaction with the treatment, consisting of 12 questions scored 1 to 5 by the patient.
Radiographic Analysis | up to 2 years
  Post-operative radiographs of the implant are analysed to identify locations and sizes of radiolucencies, indicative of poor fixation. The size, location and progression of radiolucencies is monitored. Smaller, non-progressive radiolucencies are preferred.

CONTACTS AND LOCATIONS:
Overall Officials: Atul Kamath, MD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No